CLINICAL TRIAL: NCT05681598
Title: Diagnosis and Treatment With Hydroxyurea of Sickle Cell Anemia in Democratic Republic of the Congo
Brief Title: Hydroxyurea Treatment for Adult Sickle Cell Anemia Patients in Kinshasa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kinshasa (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Principal Investigator, Paul Lumbala Kabuyi, Principal investigator, University of Kinshasa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZRDC2015PR088
Record Dates: First submitted 2022-10-06; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-12

CONDITIONS: Sickle-Cell Anaemia
Keywords: sickle cell anemia; hydroxyurea; adult patients; kinshasa
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hydroxyurea

STUDY DESIGN:
Intervention Model Description: all eligible patients received during the study period were included and received treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hydroxyurea treatment (Experimental): participants were treated with hydroxyurea
  Interventions: Drug: Hydroxyurea

INTERVENTIONS:
Drug: Hydroxyurea — The treatment started with a dose of 15mg/kg/day of HU. This initial dose was increased in steps of 5mg/kg/day every three months up to 35mg/kg/day or a maximal tolerated dose.

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of hydroxyurea (HU) in improving disease severity in adult patients with sickle cell anemia in Kinshasa (Democratic Republic of Congo). This study aims to:

* assess the safety and efficacy of HU treatment in the Congolese environment;
* assess the reversibility of chronic cardiac lesions. Participants will take hydroxyurea for two years. The effects of the treatment will be evaluated periodically by clinical evaluation, biological tests, and echocardiographic exploration.

DETAILED DESCRIPTION:
Sickle cell disease is common in sub-Saharan Africa, particularly in the Democratic Republic of the Congo (DRC). It is characterized by chronic hemolytic anemia with the need for transfusions, painful osteoarticular crises, and chronic organ damage, including the heart.

Hydroxyurea (HU) is a drug widely used in sickle cell patients in wealthy countries, while it is little used in poor countries with a high incidence of the disease.

This prospective study will focus on homozygous sickle cell participants, naïve to HU treatment. Participants will take HU in gradually increasing doses. They will be monitored for the possible occurrence of side effects. The effectiveness of the treatment will be evaluated according to the reduction in painful crises, and the need for blood transfusion; as well as based on biological changes and the reversibility or stabilization of cardiovascular complications.

ELIGIBILITY:
Inclusion Criteria:

* sickle cell anemia confirmed by DNA testing;
* moderate to severe clinical severity of sickle cell anemia;
* fetal hemoglobin lower than 15%.

Exclusion Criteria:

* poor compliance to follow-up consultation during the observational year
* participant already treated with HU
* pregnant women
* breastfeeding women
* congenital heart disease
* pulmonary disease

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 166 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2020-05-16 (Actual); Study Completion 2020-05-16 (Actual)

PRIMARY OUTCOMES:
changes from baseline in body mass index (BMI) to year 2 | baseline, year 1 and year 2
  weight in kilograms and height in meters will be combined to report BMI in kg/m^2. The measurements obtained after 1 year and after 2 years of treatment will be compared with the baseline.
changes from baseline in the frequency of Acute clinical events to year 2 | baseline, year 1 and year 2
  The number of vaso-occlusive crises and the number of transfusions and the number of days of hospitalization will be recorded each month and compiled to provide an annual assessment of the severity of the disease. The overall assessment will be 24 months.
changes from baseline in complete blood count to year 2 | baseline, 3, 6, 9, 12, 15, 18, 21 and 24 months
  A complete blood count will be assessed every 3 months up to 24 months of HU treatment. The values measured during the treatment will be compared to the basal values.
changes from baseline in Fetal hemoglobin to year 2 | baseline, 3, 6, 9, 12, 15, 18, 21 and 24 months
  The fetal hemoglobin rate will be measured every 3 months up to 24 months of HU treatment and its values compared to its initial value.
changes from baseline in left ventricle dilation to year 1 | baseline, 4, 8 and 12 months
  Left ventricular internal diameter in diastole (LVID), mesured by cardiac ultrasound, indexed to body surface area (cm/m²) will be measured at baseline and compared with measurements taken every 4 months, over a total period of 12 months of HU treatment.
changes from baseline in the thickness of left ventricular walls to year 1 | baseline, 4, 8 and 12 months
  The thickness of the walls of the left ventricle (interventricular septum and posterior wall of the left ventricle) expressed in "cm" were measured on echocardiography. The measurements taken every 4 months were compared to the basal measurement. The overall assessment will cover 12 months of treatment.
changes from baseline in the tricuspid regurgitation jet velocity to year 1 | baseline, 4, 8 and 12 months
  The velocity of the tricuspid regurgitation jet will be evaluated by cardiac ultrasound with continuous Doppler. A velocity greater than or equal to 2.5m/s indicates pulmonary hypertension. The measurement will be made every four months, for a total period of 12 months.
changes from baseline in the pulmonary acceleration time (PaccT) to year 1 | baseline, 4, 8 and 12 months
  In cardiac ultrasound short -axis view, with the pulsed-wave Doppler placed at the center of the trans-pulmonary valve jet, the PaccT is the time interval between the onset of ejection and the peak flow velocity (in milliseconds). Pulmonary hypertension will be diagnosed when PaccT was less than 90 milliseconds. The measurement will be made every four months, for a total period of 12 months.
Changes from baseline in E and A mitral to year 1 | baseline, 4, 8 and 12 months
  The transmitral Doppler velocities will be studied, with the pulsed-wave Doppler sample volume placed at the tips of the mitral valve leaflets from the apical four chambers view. Diastolic peaks velocity early (E) and later (A) will be recorded in cm/second. The measurements will be obtained at starting and every 4 months during a year of treatment.
Changes from baseline in E' mitral to year 1 | baseline, 4, 8 and 12 months
  The pulsed-wave tissue Doppler imaging (TDI) will be used to provide ventricular wall motion velocity measurements by positioning the sample volume at the parietal side of the mitral valve annuli. The velocity of the early diastolic wave (E') will be measured in cm/s. Baseline value and values obtained every 4 months will be recorded.
Changes from baseline in the E/E' mitral ratio to year 1 | baseline, 4, 8 and 12 months
  The calculated E/E' mitral ratio less than 8 indicates low filling pressures of the left ventricle. Baseline value and values obtained every 4 months during treatment will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Prosper Lukusa Tshilobo, Study Director — Center of human genetics. Faculty of medicine. University of Kinshasa
Locations (1):
- University of Kinshasa, Kinshasa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: No